CLINICAL TRIAL: NCT02015455
Title: Lumbar Imaging With Reporting of Epidemiology: A Pragmatic Cluster Randomized Trial
Brief Title: Trial of Inserting Prevalence Information Into Lumbar Spine Imaging Reports
Acronym: LIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mayo Clinic (Other); Henry Ford Health System (Other); Kaiser Permanente (Other); Oregon Health and Science University (Other); National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jeffrey G. Jarvik, MD, MPH, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 44083; UH3AR066795 (NIH); 1UH2AT007766-01 (NIH)
Record Dates: First submitted 2013-12-06; First posted 2013-12-19 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain; Back Pain; Lumbar Pain; Backache
Keywords: pragmatic trial; stepped-wedge design; cluster-randomized trial
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): Epidemiologic benchmarks included in lumbar imaging reports
  Interventions: Other: Epidemiologic benchmarks included in lumbar imaging reports
- Usual Care Arm (No Intervention): Clinics with typical lumbar imaging reports (no epidemiologic benchmarks included)

INTERVENTIONS:
Other: Epidemiologic benchmarks included in lumbar imaging reports — Epidemiologic benchmarks inserted into lumbar imaging reports
  Arms: Intervention Arm

SUMMARY:
The overall goal of the Lumbar Image Reporting with Epidemiology (LIRE) is to perform a large, pragmatic, cluster randomized controlled trial to determine the effectiveness of a simple, inexpensive and easy to deploy intervention - insertion of epidemiological benchmarks into lumbar spine imaging reports - at reducing subsequent tests and treatments. The investigator's main hypothesis is that for patients referred from primary care providers, inserting epidemiological evidence in lumbar spine imaging reports will reduce subsequent diagnostic and therapeutic interventions, including cross-sectional imaging (MR/CT), opioid prescriptions, spinal injections and surgery.

DETAILED DESCRIPTION:
The long-term public health significance is that a simple, inexpensive intervention has the potential to substantially reduce unnecessary and expensive care for back pain patients. Importantly, this approach could be applied to a wide range of other conditions and other diagnostic tests (e.g. other imaging tests, laboratory tests, genetic testing). If this study is positive, adding epidemiologic benchmarks to diagnostic test reporting could become the dominant paradigm for communicating all diagnostic information.

To test this hypothesis, the investigators propose to conduct a pragmatic cluster, randomized controlled trial, randomly assigning primary care clinics at four large health systems to receive either standard lumbar spine imaging reports or reports containing epidemiological benchmarks for common imaging findings. The investigators will use a novel stepped wedge randomization scheme that temporally randomizes sites, allowing within-site before/after comparisons in addition to between-site comparisons, while assuring that all sites will eventually receive the intervention. The primary outcome will be a metric of back-related intervention intensity. The primary analysis will occur at the clinic level and not the patient level.

This pragmatic trial will demonstrate both the feasibility of randomly assigning clinics within large health systems as well as the feasibility of passively collecting outcomes data up to two years after enrollment using the robust electronic medical records systems available at each health system.

ELIGIBILITY:
Inclusion Criteria:

* Imaging of lumbar spine requested by primary care provider

Exclusion Criteria:

* Age < 18years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250401 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G Jarvik, MD, MPH, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Kaiser Permanente of Northern California, Oakland, California
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Health Systems, Minneapolis, Minnesota
  - Group Health Cooperative, Seattle, Washington

REFERENCES:
- [Result] Jarvik JG, Comstock BA, James KT, Avins AL, Bresnahan BW, Deyo RA, Luetmer PH, Friedly JL, Meier EN, Cherkin DC, Gold LS, Rundell SD, Halabi SS, Kallmes DF, Tan KW, Turner JA, Kessler LG, Lavallee DC, Stephens KA, Heagerty PJ. Lumbar Imaging With Reporting Of Epidemiology (LIRE)--Protocol for a pragmatic cluster randomized trial. Contemp Clin Trials. 2015 Nov;45(Pt B):157-163. doi: 10.1016/j.cct.2015.10.003. Epub 2015 Oct 19. PMID 26493088
- [Result] Jarvik JG, Meier EN, James KT, Gold LS, Tan KW, Kessler LG, Suri P, Kallmes DF, Cherkin DC, Deyo RA, Sherman KJ, Halabi SS, Comstock BA, Luetmer PH, Avins AL, Rundell SD, Griffith B, Friedly JL, Lavallee DC, Stephens KA, Turner JA, Bresnahan BW, Heagerty PJ. The Effect of Including Benchmark Prevalence Data of Common Imaging Findings in Spine Image Reports on Health Care Utilization Among Adults Undergoing Spine Imaging: A Stepped-Wedge Randomized Clinical Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2015713. doi: 10.1001/jamanetworkopen.2020.15713. PMID 32886121
- [Derived] Gold LS, Marcum ZA, Meier EN, Turner JA, James KT, Kallmes DF, Luetmer PH, Griffith B, Sherman KJ, Friedly JL, Suri P, Deyo RA, Johnston SK, Avins AL, Heagerty PJ, Jarvik JG. Patient, Provider, and Clinic Characteristics Associated with Opioid and Non-Opioid Pain Prescriptions for Patients Receiving Low Back Imaging in Primary Care. J Am Board Fam Med. 2021 Sep-Oct;34(5):950-963. doi: 10.3122/jabfm.2021.05.210033. PMID 34535520
- [Derived] Suri P, Meier EN, Gold LS, Marcum ZA, Johnston SK, James KT, Bresnahan BW, O'Reilly M, Turner JA, Kallmes DF, Sherman KJ, Deyo RA, Luetmer PH, Avins AL, Griffith B, Heagerty PJ, Rundell SD, Jarvik JG, Friedly JL. Providing Epidemiological Data in Lumbar Spine Imaging Reports Did Not Affect Subsequent Utilization of Spine Procedures: Secondary Outcomes from a Stepped-Wedge Randomized Controlled Trial. Pain Med. 2021 Jun 4;22(6):1272-1280. doi: 10.1093/pm/pnab065. PMID 33595635
- [Derived] Marcum ZA, Gold LS, James KT, Meier EN, Turner JA, Kallmes DF, Cherkin DC, Deyo RA, Sherman KJ, Luetmer PH, Avins AL, Griffith B, Friedly JL, Suri P, Heagerty PJ, Jarvik JG. Effects of Including Epidemiologic Data in Lumbar Spine Imaging Reports on Prescribing Non-Opioid Medications for Pain. J Gen Intern Med. 2021 Aug;36(8):2237-2243. doi: 10.1007/s11606-021-06627-6. Epub 2021 Feb 8. PMID 33559061
- [Derived] Johnson KE, Neta G, Dember LM, Coronado GD, Suls J, Chambers DA, Rundell S, Smith DH, Liu B, Taplin S, Stoney CM, Farrell MM, Glasgow RE. Use of PRECIS ratings in the National Institutes of Health (NIH) Health Care Systems Research Collaboratory. Trials. 2016 Jan 16;17:32. doi: 10.1186/s13063-016-1158-y. PMID 26772801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 4 health systems if they had lumbar spine imaging ordered by a primary care provider that occurred between October 2013 and September 2016.
Pre-assignment Details: Of 250,401 enrolled participants, 238,886 met inclusion and exclusion criteria.
Units Other Than Participants: Clinics
Groups:
- Control: Participants with index imaging at a clinic prior to the randomized date at which the clinic started the intervention.
- Intervention: Participants with index imaging at a clinic on or after the randomized date at which the clinic started the intervention.
Period: Step 0 - Oct 2013 to Mar 2014
Arm/Group | Control | Intervention
Started (By pretrial design, for 1 site (21 clinics), step 0 extended through May 2014, and step 1 began June 2014.) | 48233; 98 Clinics | 0; 0 Clinics
Did Not Receive Intended Inclusion/Exclusion of Intervention Report Text | 135; 98 Clinics | 0; 0 Clinics
Completed | 48233; 98 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics
Period: Step 1 - Apr 2014 to Sep 2014
Arm/Group | Control | Intervention
Started (By pretrial design, for 1 site (21 clinics), step 0 extended through May 2014, and step 1 began June 2014.) | 24074; 79 Clinics | 6455; 19 Clinics
Did Not Receive Intended Inclusion/Exclusion of Intervention Report Text | 390; 79 Clinics | 2208; 19 Clinics
Completed | 24074; 79 Clinics | 6455; 19 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics
Period: Step 2 - Oct 2014 to Mar 2015
Arm/Group | Control | Intervention
Started | 23139; 59 Clinics | 16285; 39 Clinics
Did Not Receive Intended Inclusion/Exclusion of Intervention Report Text | 98; 59 Clinics | 1511; 39 Clinics
Completed | 23139; 59 Clinics | 16285; 39 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics
Period: Step 3 - Apr 2015 to Sep 2015
Arm/Group | Control | Intervention
Started | 14135; 39 Clinics | 27661; 59 Clinics
Did Not Receive Intended Inclusion/Exclusion of Intervention Report Text | 72; 39 Clinics | 4915; 59 Clinics
Completed | 14135; 39 Clinics | 27661; 59 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics
Period: Step 4 - Oct 2015 to Mar 2016
Arm/Group | Control | Intervention
Started | 7874; 21 Clinics | 31316; 77 Clinics
Did Not Receive Intended Inclusion/Exclusion of Intervention Report Text | 76; 21 Clinics | 3742; 77 Clinics
Completed | 7874; 21 Clinics | 31316; 77 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics
Period: Step 5 - Apr 2016 to Sep 2016
Arm/Group | Control | Intervention
Started | 0; 0 Clinics | 39714; 98 Clinics
Did Not Receive Intended Inclusion/Exclusion of Intervention Report Text | 0; 0 Clinics | 3512; 98 Clinics
Completed | 0; 0 Clinics | 39714; 98 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: These are analyzed participant who met all inclusion criteria and did not have any exclusions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 117455 | 121431 | 238886
Age, Customized [Count of Participants; unit: Participants]
  18-39 | 21237 | 22105 | 43342
  40-60 | 45032 | 44995 | 90027
  >60 | 51186 | 54331 | 105517
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Does not include 14 patients (<0.1%) with other or unknown gender.
  Participants
    number analyzed (Participants) | 117449 | 121423 | 238872
    Female | 67915 | 69458 | 137373
    Male | 49534 | 51965 | 101499
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17754 | 18475 | 36229
  Not Hispanic or Latino | 19867 | 19276 | 39143
  Unknown or Not Reported | 79834 | 83680 | 163514
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 806 | 880 | 1686
  Asian | 13311 | 13197 | 26508
  Native Hawaiian or Other Pacific Islander | 905 | 709 | 1614
  Black or African American | 11919 | 11649 | 23568
  White | 76431 | 79142 | 155573
  More than one race | 459 | 546 | 1005
  Unknown or Not Reported | 13624 | 15308 | 28932
Region of Enrollment [Number; unit: participants]
  United States | 117455 | 121431 | 238886
Site [Count of Participants; unit: Participants]
  A | 6950 | 7388 | 14338
  B | 96275 | 100729 | 197004
  C | 7846 | 7726 | 15572
  D | 6384 | 5588 | 11972
Imaging Modality [Count of Participants; unit: Participants]
  Radiograph | 93465 | 98970 | 192435
  Computed Tomography | 494 | 449 | 943
  Magnetic Resonance | 23496 | 22012 | 45508
Charlson Comorbidity Index (CCI) [Count of Participants; unit: Participants] — The index range is 0-24 with higher values representing a greater burden of disease. The following contribute to the index with values in parentheses: congestive heart failure (2), dementia (2), chronic pulmonary disease (1), rheumatologic disease (1), mild liver disease (2) or moderate to severe liver disease (4), diabetes with chronic complications (1), hemiplegia or paraplegia (2), renal disease (1), malignant cancer (2 or 6 if metastatic solid tumor), and AIDS/HIV (4). Presence of a comorbidity was obtained from diagnosis codes in the year preceding index imaging.
  Participants
    0 | 75106 | 77973 | 153079
    1 | 20675 | 21193 | 41868
    2 | 11451 | 11760 | 23211
    3 or higher | 10223 | 10505 | 20728
Imaging Finding Status [Count of Participants; unit: Participants]
  None | 27770 | 27776 | 55546
  LIRE finding without clinically important finding | 72127 | 77065 | 149192
  Clinically important finding | 17558 | 16590 | 34148
At Least One Opioid Prescription Prior to Index [Count of Participants; unit: Participants] | 32225 | 29306 | 61531
Primary Insurance at Index [Count of Participants; unit: Participants]
  Medicare | 44362 | 46479 | 90841
  Medicaid or state-subsidized | 5546 | 6510 | 12056
  Commercial | 65375 | 66368 | 131743
  VA | 117 | 131 | 248
  Self-pay | 731 | 570 | 1301
  Unknown or not reported | 1324 | 1373 | 2697
Socioeconomic Status Index (SSI) [Mean (Standard Deviation); unit: units on a scale] — Population: Does not include 6810 patients (2.7%) with unknown SSI due to missing participant address or matching geocoding information. Sites mapped participant address to FIPS code at the block-group level using geocoding software. These codes were mapped to socioeconomic indices derived from data available from the 2010 Census Summary File 1 and the American Community Survey, 2007 to 2011, 5-year estimate data. SSI ranges from 14 to 79. Higher SSI values indicate higher levels of socioeconomic status.
  units on a scale
    number analyzed (Participants) | 114231 | 117845 | 232076
    (all) | 56.79 (6.29) | 56.76 (6.56) | 56.78 (6.43)
Health Care Professional Type [Count of Participants; unit: Participants]
  MD | 105359 | 108165 | 213524
  DO | 8131 | 9157 | 17288
  Extender (eg NP, PA) | 3965 | 4109 | 8074
Healthcare Professional Specialty [Count of Participants; unit: Participants]
  Family Medicine | 56795 | 60277 | 117072
  Internal Medicine | 59684 | 60158 | 119842
  Other | 976 | 996 | 1972
Female Healthcare Professional [Count of Participants; unit: Participants] | 62840 | 62680 | 125520
Healthcare Professional Age [Mean (Standard Deviation); unit: years] — Population: Provider age was not available for the providers of 424 participants.
  years
    number analyzed (Participants) | 117217 | 121245 | 238462
    (all) | 49.42 (8.63) | 49.22 (8.71) | 49.32 (8.67)

OUTCOME MEASURES:

1. Primary Outcome: Relative Value Unit (RVU) for Spine-related Interventions
Description: Spine-related RVUs are a composite measure of back pain interventions that combine the overall intensity of resource utilization for back pain care in a single metric. Each spine-related procedure has an RVU associated with it representing the relative cost of the work and practice components of the procedure. The outcome measure includes the sum of the RVUs of inpatient and outpatient procedures in the year following index imaging. The Medicare conversion factor during the study period was approximately $35/RVU.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: spine-related RVU
Arm/Group | Control | Intervention
Number analyzed (Participants) | 117455 | 121431
spine-related RVU | 3.53 [2.68 to 5.08] | 3.56 [2.71 to 5.12]
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.54, Mixed Models Analysis; Adjusted for site, clinic size, age, sex, image modality, comorbidity, and site time trends. Random effects for clinic and provider; Percent Difference in Median = -0.7, 95% CI 2-sided [-2.9 to 1.5] — Percent difference in median of the intervention group with respect to the control group

2. Secondary Outcome: Number of Participants With Opioid Prescription Within 12 Months of Index Imaging
Description: An indicator of one or more opioid prescriptions from a LIRE provider (a provider who ordered index imaging for one or more participants in the LIRE Trial) within 12 months of index imaging as reported in the health system medical record.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 117455 | 121431
Participants | 46220 | 41205
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.04, Mixed Models Analysis — A p-value <0.05 was considered significant; Adjusted for site, clinic size, age, sex, image modality, comorbidity, prior opioid use, site time trends. Random effects for clinic and provider; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.91 to 1.00] — Odds ratio is for the intervention group with respect to the control group

3. Secondary Outcome: Number of Participants With Opioid Prescription Within 90 Days of Index Imaging
Description: An indicator of one or more opioid prescriptions from a LIRE provider (a provider who ordered index imaging for one or more participants in the LIRE Trial) within 90 days of index imaging as reported in the health system medical record.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 117455 | 121431
Participants | 37322 | 32873
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.02, Mixed Models Analysis — The p-value is not adjusted for multiple comparisons; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.90 to 0.99] — Odds ratio is for the intervention group with respect to the control group

4. Secondary Outcome: Number of Participants With an Opioid Prescription Within 30 Days of Index Imaging
Description: An indicator of one or more opioid prescriptions from a LIRE provider (a provider who ordered index imaging for one or more participants in the LIRE Trial) within 30 days of index imaging as reported in the health system medical record.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 117455 | 121431
Participants | 31035 | 27165
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.02, Mixed Models Analysis — The p-value is not adjusted for multiple comparisons; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.91 to 0.99] — Odds ratio is for the intervention group with respect to the control group

5. Secondary Outcome: Number of Participants With Cross-sectional Imaging Within 12 Months of Plain Film Index Imaging
Description: An indicator of one or more instances of cross-sectional imaging (MRI or CT) within 12 months of plain film index imaging. Participants with cross-sectional index imaging are excluded.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Control: Participants with plain film index imaging at a clinic prior to the randomized date at which the clinic started the intervention.
- Intervention: Participants with plain film index imaging at a clinic on or after the randomized date at which the clinic started the intervention.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 93465 | 98970
Participants | 18179 | 19069

6. Secondary Outcome: Number of Participants With Cross-sectional Imaging Within 90 Days of Plain Film Index Imaging
Description: An indicator of one or more instances of cross-sectional imaging (MRI or CT) within 90 days of plain film index imaging. Participants with cross-sectional index imaging are excluded.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 93465 | 98970
Participants | 12228 | 13099

7. Secondary Outcome: Back-pain Related Estimated Payer Costs
Description: Payer costs were not evaluated due to funding constraints.
Time Frame: 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants With Spine Surgery Within 18 Month of Index Imaging
Description: An indicator or one or more spine surgeries within 18 months of index imaging. Spine surgery includes decompression surgery, spinal fusion or proxies for spine fusion, or other surgeries involving the lumbar, sacral, or thoracic spine.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 117455 | 121431
Participants | 3753 | 3785
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.74, Mixed Models Analysis — Statistical significance defined as P<0.05; Adjusted for site, clinic size, age, sex, image modality, comorbidity, site time trends. Random effects for clinic and provider; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.91 to 1.07] — Odds ratio is for the intervention group with respect to the control group

9. Secondary Outcome: Relative Value Unit (RVU) for Spine-related Interventions at 24 Months
Description: 24-month outcomes were not evaluated due to funding constraints
Time Frame: 24 months
Reporting Status: Not Posted

10. Secondary Outcome: Opioid Prescriptions at 24 Months
Description: 24-month outcomes were not evaluated due to funding constraints
Time Frame: 24 months
Reporting Status: Not Posted

11. Secondary Outcome: Cross-sectional Imaging at 24 Months
Description: 24-month outcomes were not evaluated due to funding constraints
Time Frame: 24 months
Reporting Status: Not Posted

12. Secondary Outcome: Back-pain Related Estimated Payer Costs at 24 Months
Description: 24-month outcomes were not evaluated due to funding constraints
Time Frame: 24 months
Reporting Status: Not Posted

13. Secondary Outcome: Spine- Related Surgical Interventions
Description: 24-month outcomes were not evaluated due to funding constraints
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse events for this trial were all-cause mortality within 6 months of index imaging and emergency department visit (yes/no) within 90 days of index imaging.
Description: Emergency department visit within 90 days of index imaging is reported in the serious adverse event section. The outcome was captured through the health system medical records.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 958/117455 | 953/121431
Serious Adverse Events (participants affected / at risk) | 12885/117455 | 13289/121431
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=117455) | Intervention (N=121431)
Emergency Department visit within 90 days of index imaging (General disorders) | 12885 (12885) | 13289 (13289) — Emergency Department visits were identified in the health systems' medical records.

LIMITATIONS AND CAVEATS:
Opioid prescribing decreased in the United States during our study. Although we made multiple efforts to account for this potential confounding in our modeling, residual confounding may exist. We did not collect patient-reported outcomes (PRO), so we cannot comment on outcomes such as functional status, pain, or psychosocial functioning. The decision not to collect PRO data was deliberate, based on the recognition that it could jeopardize the feasibility of this large pragmatic trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT02015455/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT02015455/SAP_001.pdf